CLINICAL TRIAL: NCT01627938
Title: A Phase II Proof of Concept Study Evaluating the Reduction of Mitoxantrone-induced Cardiotoxicity and Neurological Outcome in the Combined Use of Mitoxantrone and Dexrazoxane (Cardioxane®) in Multiple Sclerosis (MSCardioPro)
Brief Title: Study to Evaluate the Reduction of Cardiac Problems in Multiple Sclerosis Patients With Mitoxantrone and Dexrazoxane in Combination
Acronym: MSCardioPro
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. Andrew Chan (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Andrew Chan, Principal Investigator, Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RUB001CarMS; 2010-018508-95 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-26 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Mitoxantrone; Dexrazoxane; Cardioxane; cardiotoxicity; cardiac toxicity; cardiotoxic side effects; cardiac MRI; cranial MRI; LVEF; neurological outcome
MeSH Terms: conditions — Multiple Sclerosis; Cardiotoxicity | interventions — Dexrazoxane; Mitoxantrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexrazoxane (DRZ) plus Mitoxantrone (MX) (Experimental): DRZ (600 mg/m2) : MX (12 mg/m2) ratio 50:1
  Interventions: Drug: Dexrazoxane (DRZ) plus Mitoxantrone (MX)
- Placebo plus Mitoxantrone (MX) (Placebo Comparator): Placebo + MX (12 mg/m2)
  Interventions: Drug: Placebo plus Mitoxantrone (MX)

INTERVENTIONS:
Drug: Dexrazoxane (DRZ) plus Mitoxantrone (MX) — Dosage: DRZ (600 mg/m2) : MX (12 mg/m2) ratio 50:1 DRZ infusion / MX infusion once every three months over a period of 12 months, i.e. 5 infusions
  Other Names: Cardioxane® (Dexrazoxane); Ralenova® (Mitoxantrone)
  Arms: Dexrazoxane (DRZ) plus Mitoxantrone (MX)
Drug: Placebo plus Mitoxantrone (MX) — MX Dosage: 12mg/m2 Placebo infusion / MX infusion once every three months over a period of 12 months, i.e. 5 infusions
  Other Names: Ralenova ® (Mitoxantrone)
  Arms: Placebo plus Mitoxantrone (MX)

SUMMARY:
This study will primarily address the question whether the combination of Mitoxantrone therapy with dexrazoxane can reduce cardiotoxic side effects in the treatment of Multiple Sclerosis patients in comparison to Mitoxantrone monotherapy.

DETAILED DESCRIPTION:
It is designed to provide clinical and paraclinical efficacy and safety data for dexrazoxane in Mitoxantrone treatment of Multiple Sclerosis in order to investigate the possible positive influence of dexrazoxane on cardiac function of Mitoxantrone-affected myocardial tissue and on the possible augmented clinical efficacy of Mitoxantrone in combination with dexrazoxane on neurological outcome parameters. The incidence of cardiotoxicity during combined Mitoxantrone/dexrazoxane treatment will be investigated and compared to the standard Mitoxantrone-treatment without dexrazoxane.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Male or female subject is 18 years of age to 55 years of age
* Subject must have one of the below mentioned confirmed diagnoses of Multiple Sclerosis: RRMS or CPMS according to rev. McDonald Criteria (2005)
* If female of childbearing potential: Will to practice reliable birth control measures during study treatment and for at least 6 months after completion of study medication; not lactating or pregnant; and has a documented negative pregnancy test result within 72 hours prior to study medication administration. Male study participants: Will to practice reliable birth control measures during study treatment and for at least 6 months after completion of study medication
* Subject is willing to participate in the study, follow protocol study treatment regimen, and comply with all planned assessments
* Mitoxantrone treatment indication is given according to current guidelines:

  * Relapsing progressive or secondary progressive MS with/without superimposed relapses
  * EDSS 3-6; EDSS deterioration ≥1 point over last 18 months or 2 relapses
  * non-response or non-tolerability of pre-treatment
* ≥ 48 mg/m² BSA MX dose received up to baseline visit as lifetime dosage before study entry. If the patient is under regular ongoing MX treatment, the infusion interval of 3 months must be obtained (see exclusion criteria)

Exclusion Criteria:

* Concomitant clinically suspected or confirmed neurologic disorder at study entry that may interfere with the evaluation in this protocol [i.e. EDSS, MSFC, MEP or MRI measurements]
* Pre-Treatment with DRZ or immunosuppressive drugs of the anthracycline family with cardiotoxic potential other than MX prior to study enrollment
* Last Treatment with MX within the past 84 days prior to study enrollment (regular 3-monthly intervals must be obtained)
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive HCG laboratory test (>5 mIU/ml)
* Unwillingness to perform adequate contraception
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Subjects unable or unwilling to adhere to the study-designated procedures and restrictions
* Patients not able to perform cardiac/neurological investigations including MRI, e.g. hypersensitivity to MRI contrast agent
* Other known contraindication for DRZ or MX according to current labelling
* Subject has a pre-existing cardiac disease interfering with left ventricular ejection fraction, i.e. cardiac insufficience for different reasons (resulting from prior cardial conditions such as myocardial infarction, myocarditis)
* Routine co-administration of cortisone-pulse therapy (other than for treatment of relapses), intrathecal triamcinolone-therapy or other off-label/ investigational agents (e.g. fampridine, aminopyridine)
* History of malignancy in the past 5 years (excluding localized basal cell carcinoma of the skin)
* Pre-Treatment with other immunosuppressive drugs (azathioprine, methotrexate, mycophenolate, cyclophosphamide) within the past 3 months
* Pre-Treatment with monoclonal antibodies (natalizumab, rituximab) within the past 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Changes in LVEF in the different treatment arms by cardiac MRI | Baseline to month 12
  Assessment of cardiac function by measurement of LVEF in mitoxantrone plus dexrazoxane treatment arm versus mitoxantrone plus placebo treatment arm by cardiac MRI

SECONDARY OUTCOMES:
Changes in LVEF by transthoracic echocardiography and determination of cardiac side effects by ECG and by measurement of CK-MB, Troponin and BNP in mitoxantrone plus dexrazoxane versus mitoxantrone plus placebo treatment arms | Baseline and month 3,6,9,12, 24
  Assessment of cardiac function by measurement of LVEF by transthoracic echocardiography, by determination of cardiac side effects by ECG and by measurement of CK-MB, Troponin and BNP in mitoxantrone plus dexrazoxane treatment arm versus mitoxantrone plus placebo treatment arm
Determination of EDSS and relapse rate in mitoxantrone plus dexrazoxane treatment arm versus mitoxantrone plus placebo treatment arm | Baseline and month 3,6,9,12 and 24
  Comparison of clinical efficacy of mitoxantrone plus dexrazoxane treatment versus mitoxantrone plus placebo treatment on neurological outcome parameters by means of EDSS and relapse rate
Cumulative number of active lesions by cMRI | Day1 and month 12
LVEF in 3D-echocardiography vs. LVEF in cardiac MRI | Baseline and month 12
Clinical efficacy of DRZ+MX vs. MX monotherapy by MSFC | Baseline and month 3,6,9,12 and 24
Quality of Life by SF-36 questionnaire | Baseline and month 3,6,9 and month 12
Changes in magnetic evoked potentials: prolongation of TMCT+CMCT, potential configuration | Baseline and month 3,6,9 and month 12
Annual brain atrophy rates in cMRI | Day 1 and month 12
Changes in transcranial sonography (abnormal iron deposition AID). AID in cMRI. Comparison of both methods | Baseline and month 12
Analysis of ABD transporter gene polymorphisms as predictor of therapy response and side effect profile via TaqMan PCR | Baseline and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chan, PD Dr., Principal Investigator — Department of Neurology, St. Josef-Hospital Bochum, Ruhr-University Bochum
Locations (1):
- Department of Neurology, St. Josef-Hospital, Ruhr-University Bochum, Bochum, Germany

REFERENCES:
- [Background] Flachenecker P, Meissner H. Fatigue in multiple sclerosis presenting as acute relapse: subjective and objective assessment. Mult Scler. 2008 Mar;14(2):274-7. doi: 10.1177/1352458507082480. PMID 18337428
- [Background] Morrissey SP, Le Page E, Edan G. Mitoxantrone in the treatment of multiple sclerosis. Int MS J. 2005 Nov;12(3):74-87. PMID 16417821
- [Background] Rieckmann P, Toyka KV, Bassetti C, Beer K, Beer S, Buettner U, Chofflon M, Gotschi-Fuchs M, Hess K, Kappos L, Kesselring J, Goebels N, Ludin HP, Mattle H, Schluep M, Vaney C, Baumhackl U, Berger T, Deisenhammer F, Fazekas F, Freimuller M, Kollegger H, Kristoferitsch W, Lassmann H, Markut H, Strasser-Fuchs S, Vass K, Altenkirch H, Bamborschke S, Baum K, Benecke R, Bruck W, Dommasch D, Elias WG, Gass A, Gehlen W, Haas J, Haferkamp G, Hanefeld F, Hartung HP, Heesen C, Heidenreich F, Heitmann R, Hemmer B, Hense T, Hohlfeld R, Janzen RW, Japp G, Jung S, Jugelt E, Koehler J, Kolmel W, Konig N, Lowitzsch K, Manegold U, Melms A, Mertin J, Oschmann P, Petereit HF, Pette M, Pohlau D, Pohl D, Poser S, Sailer M, Schmidt S, Schock G, Schulz M, Schwarz S, Seidel D, Sommer N, Stangel M, Stark E, Steinbrecher A, Tumani H, Voltz R, Weber F, Weinrich W, Weissert R, Wiendl H, Wietholter H, Wildemann U, Zettl UK, Zipp F, Zschenderlein R, Izquierdo G, Kirjazovas A, Packauskas L, Miller D, Koncan Vracko B, Millers A, Orologas A, Panellus M, Sindic CJ, Bratic M, Svraka A, Vella NR, Stelmasiak Z, Selmaj K, Bartosik-Psujik H, Mitosek-Szewczyk K, Belniak E, Mochecka A, Bayas A, Chan A, Flachenecker P, Gold R, Kallmann B, Leussink V, Maurer M, Ruprecht K, Stoll G, Weilbach FX; Multiple Sclerosis Therapy Consensus Group. Escalating immunotherapy of multiple sclerosis--new aspects and practical application. J Neurol. 2004 Nov;251(11):1329-39. doi: 10.1007/s00415-004-0537-6. PMID 15592728
- [Background] Spindler M, Weilbach F, Beer M, Sandstede J, Kostler H, Strotmann J, Voelker W, Hahn D, Ertl G, Gold R. Non-invasive functional and biochemical assessment of mitoxantrone cardiotoxicity in patients with multiple sclerosis. J Cardiovasc Pharmacol. 2003 Nov;42(5):680-7. doi: 10.1097/00005344-200311000-00015. PMID 14576518
- [Background] Weilbach FX, Chan A, Toyka KV, Gold R. The cardioprotector dexrazoxane augments therapeutic efficacy of mitoxantrone in experimental autoimmune encephalomyelitis. Clin Exp Immunol. 2004 Jan;135(1):49-55. doi: 10.1111/j.1365-2249.2004.02344.x. PMID 14678264
- [Background] Bernitsas E, Wei W, Mikol DD. Suppression of mitoxantrone cardiotoxicity in multiple sclerosis patients by dexrazoxane. Ann Neurol. 2006 Jan;59(1):206-9. doi: 10.1002/ana.20747. PMID 16374818
- [Background] Cotte S, von Ahsen N, Kruse N, Huber B, Winkelmann A, Zettl UK, Starck M, Konig N, Tellez N, Dorr J, Paul F, Zipp F, Luhder F, Koepsell H, Pannek H, Montalban X, Gold R, Chan A. ABC-transporter gene-polymorphisms are potential pharmacogenetic markers for mitoxantrone response in multiple sclerosis. Brain. 2009 Sep;132(Pt 9):2517-30. doi: 10.1093/brain/awp164. Epub 2009 Jul 15. PMID 19605531
- [Background] Dorr J, Bitsch A, Schmailzl KJ, Chan A, von Ahsen N, Hummel M, Varon R, Lill CM, Vogel HP, Zipp F, Paul F. Severe cardiac failure in a patient with multiple sclerosis following low-dose mitoxantrone treatment. Neurology. 2009 Sep 22;73(12):991-3. doi: 10.1212/WNL.0b013e3181b878f6. No abstract available. PMID 19770476
- [Background] Hartung HP, Gonsette R, Konig N, Kwiecinski H, Guseo A, Morrissey SP, Krapf H, Zwingers T; Mitoxantrone in Multiple Sclerosis Study Group (MIMS). Mitoxantrone in progressive multiple sclerosis: a placebo-controlled, double-blind, randomised, multicentre trial. Lancet. 2002 Dec 21-28;360(9350):2018-25. doi: 10.1016/S0140-6736(02)12023-X. PMID 12504397